CLINICAL TRIAL: NCT00883116
Title: A Phase III, Open Label, Randomized, 2 Arm Study of Ixabepilone Administered Every 21 Days Versus Paclitaxel or Doxorubicin Administered Every 21 Days in Women With Advanced Endometrial Cancer Who Have Previously Been Treated With Chemotherapy
Brief Title: A Study of Ixabepilone as Second-line Therapy for Locally Advanced, Recurrent, or Metastatic Endometrial Cancer
Acronym: IXAMPLE2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis results showed that ixabepilone did not improve survival compared with control chemotherapies.
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-196; 2008-007167-16
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ixabepilone; Doxorubicin; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ixabepilone, 40 mg/m^2, intravenously (IV) (Experimental): Participants received ixabepilone, 40 mg/m^2, given IV over 3 hours every 21 days until unacceptable toxicity or disease progression
  Interventions: Drug: Ixabepilone
- Control chemotherapy (Paclitaxel or Doxorubicin) (Active Comparator): Participants received either paclitaxel, 175 mg/m^2 given IV over 3 hours, or per institutional guidelines but not exceeding 3 hours, every 21 days until disease progression or unacceptable toxicity or doxorubicin, 60 mg/m^2 given IV per institutional guidelines every 21 days, depending on the prior therapy received, until disease progression, unacceptable toxicity, or cumulative dose of 500 mg/m^2.
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ixabepilone
  Other Names: Ixempra; BMS-247550
  Arms: Ixabepilone, 40 mg/m^2, intravenously (IV)
Drug: Doxorubicin
  Other Names: Adriamycin PFS/RDF; Adriacin; Adriblastina; Adriablastine; Adrimedac; DOXO-CELL; Doxolem; Doxorubin; Farmiblastina; Rubex
  Arms: Control chemotherapy (Paclitaxel or Doxorubicin)
Drug: Paclitaxel
  Other Names: Taxol; Anzatax; Asotax; Bristaxol Praxel; Taxol Konzentrat; F1-106
  Arms: Control chemotherapy (Paclitaxel or Doxorubicin)

SUMMARY:
The primary purpose of this study is to investigate whether administration of ixabepilone results in superior outcome as assessed by overall survival compared with that achieved with standard chemotherapy (paclitaxel or doxorubicin) in women with advanced endometrial cancer that has progressed following first-line chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria

* Women aged 18 years and older
* Histologic or cytologic diagnosis of endometrial carcinoma
* Evidence that the cancer is advanced, recurrent, or metastatic and not curable by local measures, such as surgery or radiation.
* Karnofsky performance status >=70
* Measurable or nonmeasurable disease that has progressed since last treatment.

  * If only disease is confined to a solitary lesion, its neoplastic nature must be confirmed by histology or cytology.
  * Disease in a previously irradiated field is acceptable as the only site of measurable disease only if there has been clear progression since completion of radiotherapy.
* All therapy directed at endometrial cancer must be discontinued 21 days prior to start of treatment, except for hormonal therapy which must be discontinued at least 1 week prior to start of study treatment. Concurrent administration of hormone replacement therapy is allowed.
* Prior therapy: Participants must have failed 1 prior platinum-based chemotherapeutic regimen for endometrial cancer. May have received 2 prior chemotherapy regimens if 1 regimen was given for stage I or II disease. May have received any number of prior non-cytotoxic regimens such as monoclonal antibodies, cytokines, signal transduction inhibitors, or hormonal therapy. Previous radiation therapy is allowed.

Key Exclusion Criteria

* Carcinosarcoma (malignant mixed mullerian tumor)
* Endometrial leiomyosarcoma and endometrial stromal sarcomas
* Participants who received no prior chemotherapy for endometrial cancer or ≥2 prior chemotherapy regimens (exceptions defined in protocol)
* Known brain metastases
* Receipt of prior ixabepilone therapy
* Concurrent active infection requiring antibiotics or other therapy
* Concurrent unstable disease or other debilitating illness, such as congestive heart failure, unstable angina, myocardial infarction, or other cardiac disease that could jeopardize participation, within the last 6 months
* For participants whose prior therapy did not include an anthracycline and therefore may be randomized to doxorubicin, left ventricular ejection fraction <50% as measured by multigated radionuclide angiography or echocardiography
* History of malignancy, except nonmelanoma skin cancer, carcinoma in situ of the cervix, or carcinoma in situ of the breast, within the last 5 years that has not been treated with chemotherapy
* Known human immunodeficiency viral infection
* Psychiatric disorders or other conditions rendering the participant incapable of complying with protocol requirements
* Absolute neutrophil count <1500/mm^3
* Platelets <100,000/mm^3
* Hemoglobin <9 g/dL
* Total bilirubin >1.5*upper limit of normal (ULN), except for those with Gilbert's disease
* Aspartate aminotransferase or alanine aminotransferase >2.5*ULN
* Serum creatinine >1.5*ULN
* Grade ≥2 neuropathy (sensory or motor)
* No concurrent therapy (chemotherapy, hormonal, or investigational) directed at endometrial cancer during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (89):
- United States (28):
  - University Of South Alabama, Mobile, Alabama
  - Rocky Mountain Gynecologic Oncology, Englewood, Colorado
  - Peter E. Schwartz, Md, New Haven, Connecticut
  - Hematology Oncology, P.C., Stamford, Connecticut
  - Gynecologic Oncology Assoc.,Inc, Hollywood, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Georgia Health Science University, Augusta, Georgia
  - Sudarshan K. Sharma, Md, Hinsdale, Illinois
  - Central Dupage Hospital Cancer Center, Warrenville, Illinois
  - St. Vincent Hospital And Health Care Center, Inc., Indianapolis, Indiana
  - Hematology And Oncology Specialists, Llc, Marrero, Louisiana
  - Women'S Health Specialists, Rockville, Maryland
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - University Of Minnesota, Minneapolis, Minnesota
  - Saint Dominic's Gynecologic Oncology, Jackson, Mississippi
  - Matthew A Powell, Md, St Louis, Missouri
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Peggy And Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Magee-Womens Hospital Of Upmc Laboratory, Pittsburgh, Pennsylvania
  - Women & Infants Hospital Of Ri, Providence, Rhode Island
  - Cancer Centers Of The Carolinas, Greenville, South Carolina
  - Tennessee Gynecologic Oncology Group, Llc, Chattanooga, Tennessee
  - University Of Virginia, Charlottesville, Virginia
- Argentina (3):
  - Local Institution, La Rioja, La Rioja Province
  - Local Institution, Salta, Salta Province
  - Local Institution, Rosario, Santa Fe Province
- Australia (2):
  - Local Institution, Milton, Queensland
  - Local Institution, East Bentleigh, Victoria
- Belgium (2):
  - Local Institution, Ghent
  - Local Institution, Leuven
- Brazil (4):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, Jaú, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (7):
  - Local Institution, Calgary, Alberta
  - Local Institution, Surrey, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, Toronto, Ontario
  - Local Institution, Fleurimont, Quebec
  - Local Institution, Montreal, Quebec
- Czechia (2):
  - Local Institution, Brno
  - Local Institution, Hradec Králové
- Denmark (3):
  - Local Institution, Copenhagen
  - Local Institution, Herlev
  - Local Institution, Odense C
- France (4):
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Saint-Herblain
  - Local Institution, Villejuif
- Local Institution, Athens, Greece
- Hungary (2):
  - Local Institution, Budapest
  - Local Institution, Miskolc
- Italy (6):
  - Local Institution, Brescia
  - Local Institution, Campobasso
  - Local Institution, Meldola (fc)
  - Local Institution, Milan
  - Local Institution, Monza
  - Local Institution, Roma
- Mexico (5):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Mexico City
  - Local Institution, Tlalpan, Mexico City
- Norway (2):
  - Local Institution, Bergen
  - Local Institution, Oslo
- Local Institution, Lima, Lima Province, Peru
- Russia (5):
  - Local Institution, Ivanovo
  - Local Institution, Moscow
  - Local Institution, Obninsk
  - Local Institution, Saint Pertersburg
  - Local Institution, Saint Petersburg
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Valencia
- Sweden (5):
  - Local Institution, Gothenburg
  - Local Institution, Linköping
  - Local Institution, Stockholm
  - Local Institution, Umeå
  - Local Institution, Uppsala
- United Kingdom (4):
  - Local Institution, Bristol, Avon
  - Local Institution, Glasgow, Dumfries & Galloway
  - Local Institution, Nottingham, Nottinghamshire
  - Local Institution, Leeds, Yorkshire

REFERENCES:
- [Derived] McMeekin S, Dizon D, Barter J, Scambia G, Manzyuk L, Lisyanskaya A, Oaknin A, Ringuette S, Mukhopadhyay P, Rosenberg J, Vergote I. Phase III randomized trial of second-line ixabepilone versus paclitaxel or doxorubicin in women with advanced endometrial cancer. Gynecol Oncol. 2015 Jul;138(1):18-23. doi: 10.1016/j.ygyno.2015.04.026. Epub 2015 Apr 26. PMID 25925990
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 551 participants enrolled. 496 randomized (248 ixabepilone, 248 control); 487 received treatment (248 ixabepilone, 239 to control). Reasons not treated include 1 no longer met study criteria, 1 withdrew consent, 1 condition worsened, and 6 non-specified.
Groups:
- Ixabepilone, 40 mg/m^2, IV: Participants received ixabepilone, 40 mg/m^2, given intravenously (IV) over 3 hours every 21 days until unacceptable toxicity or disease progression
- Control Chemotherapy: Participants received either paclitaxel, 175 mg/m^2 given IV over 3 hours, or per institutional guidelines but not exceeding 3 hours, every 21 days until disease progression or unacceptable toxicity or doxorubicin, 60 mg/m^2 given IV per institutional guidelines every 21 days, depending on the prior therapy received, until disease progression, unacceptable toxicity, or cumulative dose of 500 mg/m^2.
Period: Overall Study
Arm/Group | Ixabepilone, 40 mg/m^2, IV | Control Chemotherapy
Started | 248 | 248
Received Treatment | 248 | 239
Completed | 39 | 29
Not Completed | 209 | 219
Not completed — Adverse event unrelated to study drug | 5 | 10
Not completed — Death | 6 | 2
Not completed — Disease progression | 130 | 128
Not completed — Lost to Follow-up | 0 | 1
Not completed — Maximum clinical benefit | 13 | 46
Not completed — Not identified | 3 | 6
Not completed — Study drug toxicity | 36 | 16
Not completed — Withdrawal by Subject | 14 | 8
Not completed — No longer meets study criteria | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analyses are for randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 40 mg/m^2, IV | Control Chemotherapy | Total
Number analyzed (Participants) | 248 | 248 | 496
Age, Continuous [Median (Full Range); unit: Years] | 64.0 [39.0 to 86.0] | 64.0 [33.0 to 88.0] | 64.0 [33.0 to 88.0]
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 126 | 139 | 265
  65 years and older | 122 | 109 | 231
  Younger than 50 years | 14 | 18 | 32
  50 years and older | 234 | 230 | 464
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 248 | 248 | 496
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 215 | 213 | 428
  Black or African American | 12 | 18 | 30
  Asian | 6 | 5 | 11
  Other | 12 | 12 | 24
  American Indian or Alaska Native | 3 | 0 | 3
Karnofsky Performance Scale Index Status [Number; unit: Participants] — This scale classifies patients by functional impairment. The lower the Karnofsky score, the more impaired the patient is. 100=No complaints; 90=Normal activity; 80=Normal activity with effort; 70=Cares for self but unable to carry on normal activity or to do active work; 60=Requires occasional assistance, but is able to care for most of his personal needs; 50=Requires considerable assistance; 40=Disabled; requires special care; 30=Severely disabled hospitalization indicated; 20=Very sick; hospital admission necessary; 10=Fatal processes progressing rapidly; 0=Death.
  Participants
    100 | 86 | 86 | 172
    90 | 95 | 79 | 174
    80 | 48 | 64 | 112
    70 | 19 | 16 | 35
    <70 | 0 | 2 | 2
    Not reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Survival was defined as the time from the date of randomization until the date of death. If the patient did not die, OS was censored on the last date he or she was known to be alive.
Time Frame: Date of randomization to date of death or last date censored to up to approximately 26 months
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Control With Chemotherapy (Paclitaxel or Doxorubicin): Participants received paclitaxel, 175 mg/m^2, given IV over 3 hours, or per institutional guidelines but not exceeding 3 hours, every 21 days until disease progression or unacceptable toxicity or doxorubicin, 60 mg/m^2, given IV per institutional guidelines every 21 days, depending on the prior therapy received, until disease progression, unacceptable toxicity, or cumulative dose of 500 mg/m^2.
Arm/Group | Ixabepilone, 40 mg/m^2, Intravenously (IV) | Control With Chemotherapy (Paclitaxel or Doxorubicin)
Number analyzed (Participants) | 248 | 248
Months | 10.9 [8.5 to 12.7] | 12.3 [10.7 to 15.4]
Statistical Analysis 1: Comparison: Ixabepilone, 40 mg/m^2, Intravenously (IV) vs Control With Chemotherapy (Paclitaxel or Doxorubicin); Test type: Superiority or Other; p = 0.0397, Log Rank; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [1.0 to 1.7]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the date of documented disease progression. Patients who died without a reported prior progression were considered to have progressed on the date of their death. Those who did not progress or die were censored on the date of their last tumor assessment. Participants who did not have any on-study tumor assessments were censored on the date they were randomized. Measurable disease was present if the patient had 1 or more measurable lesions.
Time Frame: Date of randomization to date of disease progression or death (or date of last tumor assessment for those who did not die or progress) up to approximately 22 months
Population: All participants with measurable disease at randomization
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Control With Chemotherapy (Paclitaxel or Doxorubicin): Participants received either paclitaxel, 175 mg/m^2 given IV over 3 hours, or per institutional guidelines but not exceeding 3 hours, every 21 days until disease progression or unacceptable toxicity or doxorubicin, 60 mg/m^2 given IV per institutional guidelines every 21 days, depending on the prior therapy received, until disease progression, unacceptable toxicity, or cumulative dose of 500 mg/m^2.
Arm/Group | Ixabepilone, 40 mg/m^2, Intravenously (IV) | Control With Chemotherapy (Paclitaxel or Doxorubicin)
Number analyzed (Participants) | 223 | 223
Months | 3.4 [2.8 to 4.2] | 4.0 [2.7 to 4.3]
Statistical Analysis 1: Comparison: Ixabepilone, 40 mg/m^2, Intravenously (IV) vs Control With Chemotherapy (Paclitaxel or Doxorubicin); Test type: Superiority or Other; p = 0.8011, Log Rank; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.8 to 1.3]

3. Secondary Outcome: Best Overall Response Rate
Description: Best overall response rate was defined as the number of participants whose best response was either partial response (PR) or complete response (CR) divided by the number of participants in the treatment group. Overall tumor response was based on an integration of the evaluation of target, nontarget, and new lesions. CR=Disappearance of all clinical and radiologic evidence of target lesions. PR=At least 30% reduction in the sum of diameters of all target lesions; taking as reference the baseline study measurement. Changes in tumor measurements need not be confirmed by repeat measurements performed after the criteria for response were first met.
Time Frame: Date of randomization and every 6 weeks to end of treatment (9 cycles, or approximately Day 189)
Population: All randomized participants with measurable disease
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ixabepilone, 40 mg/m^2, Intravenously (IV) | Control With Chemotherapy (Paclitaxel or Doxorubicin)
Number analyzed (Participants) | 223 | 223
Percentage of participants | 15.2 [10.8 to 20.6] | 15.7 [11.2 to 21.1]

4. Secondary Outcome: Number of Participants With a Serious Adverse Event (SAE), an SAE Related to Study Drug, Death as Outcome, a Peripheral Neuropathy Adverse Event (AE), a Grade 3 or Higher AE, and an AE Related to Study Drug
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related to study drug=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: From Day 1 (first dose) to 30 days past last dose (up to Day 219); 9 cycles, or 189 days + 30 days
Population: All participants who received at least 1 dose of ixabepilone
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 40 mg/m^2, Intravenously (IV) | Control With Chemotherapy (Paclitaxel or Doxorubicin)
Number analyzed (Participants) | 248 | 239
Participants
  Any SAEs | 89 | 70
  Any SAE related to study drug | 43 | 29
  Deaths | 121 | 95
  Any AE related to study drug | 223 | 215
  Any AE leading to study drug discontinuation | 49 | 37
  Any peripheral neuropathy AE | 108 | 62
  Any Grade 3 or higher AE | 160 | 148

ADVERSE EVENTS:
Time Frame: Day 1 up to 30 days post last dose of study therapy, an average of 4 years
Description: Study initiated: August 2009; Study Completion: February 2014
Groups:
- Ixabepilone, 40 mg/m^2, Intravenously (IV): Participants received ixabepilone, 40 mg/m^2, given intravenously (IV) over 3 hours every 21 days until unacceptable toxicity or disease progression
- Control With Chemotherapy (Doxorubicin, 60 mg/m^2, IV): Participants received doxorubicin, 60 mg/m^2 given intravenously (IV) per institutional guidelines every 21 days, depending on the prior therapy received, until disease progression, unacceptable toxicity, or cumulative dose of 500 mg/m^2.
- Control With Chemotherapy (Paclitaxel, 175 mg/m^2, IV): Participants received paclitaxel, 175 mg/m^2 given IV over 3 hours, or per institutional guidelines but not exceeding 3 hours, every 21 days until disease progression or unacceptable toxicity.
Arm/Group | Ixabepilone, 40 mg/m^2, Intravenously (IV) | Control With Chemotherapy (Doxorubicin, 60 mg/m^2, IV) | Control With Chemotherapy (Paclitaxel, 175 mg/m^2, IV)
Serious Adverse Events (participants affected / at risk) | 89/248 | 59/171 | 11/68
Other Adverse Events (participants affected / at risk) | 233/248 | 160/171 | 63/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 40 mg/m^2, Intravenously (IV) (N=248) | Control With Chemotherapy (Doxorubicin, 60 mg/m^2, IV) (N=171) | Control With Chemotherapy (Paclitaxel, 175 mg/m^2, IV) (N=68)
Blood creatinine increased (Investigations) | 3 | 0 | 0
Device malfunction (General disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Dyspnoea exertional (Reproductive system and breast disorders) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 10 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0
Sudden death (General disorders) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0
Inflammation (General disorders) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 7 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 4 | 0
Salmonellosis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 3 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 2
Asthenia (General disorders) | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 2 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 0
Pain (General disorders) | 1 | 0 | 1
Respiratory moniliasis (Infections and infestations) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 4 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 1
General physical health deterioration (General disorders) | 1 | 0 | 1
Infectious peritonitis (Infections and infestations) | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 1
Septic shock (Infections and infestations) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 4 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 2 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 4 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 40 mg/m^2, Intravenously (IV) (N=248) | Control With Chemotherapy (Doxorubicin, 60 mg/m^2, IV) (N=171) | Control With Chemotherapy (Paclitaxel, 175 mg/m^2, IV) (N=68)
Dizziness (Nervous system disorders) | 24 | 10 | 1
Dyspepsia (Gastrointestinal disorders) | 17 | 14 | 0
Decreased appetite (Metabolism and nutrition disorders) | 82 | 45 | 12
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 6
Neuropathy peripheral (Nervous system disorders) | 17 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 12 | 8
Anxiety (Psychiatric disorders) | 11 | 13 | 1
Dysgeusia (Nervous system disorders) | 23 | 18 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37 | 33 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 13 | 7 | 0
Leukopenia (Blood and lymphatic system disorders) | 35 | 25 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 16 | 5
Peripheral motor neuropathy (Nervous system disorders) | 12 | 2 | 5
Haemoglobin decreased (Investigations) | 13 | 11 | 3
Nausea (Gastrointestinal disorders) | 118 | 101 | 17
Peripheral sensory neuropathy (Nervous system disorders) | 79 | 10 | 29
Pyrexia (General disorders) | 17 | 22 | 4
Vaginal haemorrhage (Reproductive system and breast disorders) | 13 | 2 | 4
Weight increased (Investigations) | 3 | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 45 | 24 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 102 | 63 | 36
Asthenia (General disorders) | 39 | 24 | 11
Mucosal inflammation (General disorders) | 21 | 28 | 0
Neutropenia (Blood and lymphatic system disorders) | 58 | 68 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 12 | 2
Weight decreased (Investigations) | 48 | 28 | 3
Abdominal pain upper (Gastrointestinal disorders) | 7 | 14 | 1
Anaemia (Blood and lymphatic system disorders) | 62 | 46 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 9 | 22
Constipation (Gastrointestinal disorders) | 77 | 49 | 7
Dehydration (Metabolism and nutrition disorders) | 14 | 8 | 0
Diarrhoea (Gastrointestinal disorders) | 76 | 47 | 8
Lymphopenia (Blood and lymphatic system disorders) | 7 | 11 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 32 | 4 | 17
Stomatitis (Gastrointestinal disorders) | 16 | 18 | 1
Vomiting (Gastrointestinal disorders) | 73 | 48 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 15 | 3
Fatigue (General disorders) | 125 | 88 | 21
Headache (Nervous system disorders) | 19 | 16 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 14 | 2
Insomnia (Psychiatric disorders) | 28 | 13 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8 | 3 | 4
Oedema peripheral (General disorders) | 27 | 20 | 6
Paraesthesia (Nervous system disorders) | 10 | 3 | 5
Rash (Skin and subcutaneous tissue disorders) | 21 | 7 | 3
Urinary tract infection (Infections and infestations) | 22 | 9 | 3

LIMITATIONS AND CAVEATS:
This study was terminated per Data Monitoring Committee. Results from an interim analysis showed that there was no favorable benefit/risk ratio with ixabepilone and that ixabepilone did not improve survival compared with control chemotherapies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.